CLINICAL TRIAL: NCT02910310
Title: Introduction of a Uterine Balloon Tamponade for Postpartum Hemorrhage in Three Low Income Countries: a Stepped Wedge Cluster Randomized Trial
Brief Title: Introduction of UBT for PPH Management in Three Countries
Acronym: UBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Ministry of Health and Population, Egypt (Other Government); Alexandria University (Other); El Galaa Teaching Hospital (Other); Global Health Uganda LTD (Other); Makerere University (Other); Ministry of Health, Uganda (Other Government); Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3005
Record Dates: First submitted 2016-09-15; First posted 2016-09-22 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine Balloon Tamponade
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Uterine Balloon Tamponade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baseline period (No Intervention): The baseline period will involve data collection on study outcomes before uterine balloon tamponade (UBT) is introduced at study sites.
- Uterine balloon tamponade (Experimental): The UBT period will involve data collection on study outcomes after providers at sites are trained on UBT use and UBT is introduced into PPH management practice at study sites.
  Interventions: Other: Uterine balloon tamponade

INTERVENTIONS:
Other: Uterine balloon tamponade — An intervention consisting of inserting a condom attached to a urinary catheter into the uterus and inflating it with fluid to stop postpartum bleeding
  Arms: Uterine balloon tamponade

SUMMARY:
This study is a prospective, systematic evaluation to assess the effectiveness and safety of introduction of UBT into PPH care at secondary level and district hospitals in 3 low-resource countries. The first component of the evaluation is a prospective stepped wedge cluster randomized design to assess the potential reduction in PPH-related mortality and invasive procedures (blood transfusion, arterial ligation, hysterectomy and uterine arterial embolization) for PPH performed at participating facilities following introduction of UBT. The second component is a nested cohort analysis to assess the safety and acceptability of UBT among women diagnosed with PPH.

DETAILED DESCRIPTION:
To assess the effectiveness of introduction of the UBT, a stepped wedge cluster randomized design will be employed to monitor maternal health outcomes among vaginal deliveries occurring at all participating facilities during the study phases described below:

Baseline phase: A baseline phase will be conducted in all participating sites before training and introduction of the UBT for PPH management. This phase will consist of prospective data collection to establish the baseline rates of key study outcomes.

Step 1 intervention phase: In this phase, participating sites will be randomized such that half will receive training on use of the UBT for PPH management with subsequent introduction into their standard practice and half will continue data collection without UBT introduction.

Step 2 intervention phase: In this phase, the remaining sites will receive training on use of the UBT for PPH management with subsequent introduction into their standard practice. During this phase, all participating sites will continue data collection to document study outcomes and all will be using UBT in their standard practice.

To assess the safety and acceptability of the use of UBT for PPH management, a nested cohort analysis will be done among women diagnosed with PPH during the stepped wedge trial. The investigators will assess the rates of treatment of postpartum infection and examine acceptability of care provided among the following two cohorts of women:

UBT group: All women diagnosed with PPH following a vaginal delivery and who have an attempted UBT placement (including successful or unsuccessful placements).

No-UBT group: All women diagnosed with PPH following a vaginal delivery that do not have an attempted UBT placement.

ELIGIBILITY:
Eligibility for stepped wedge trial:

Inclusion Criteria:

* Vaginal delivery at participating facility or referred to participating facility for PPH after vaginal delivery elsewhere

Exclusion Criteria:

* Delivery via Cesarean section
* Transferred to another facility before delivery
* Transferred to the participating facility after vaginal delivery elsewhere but died before arrival

Eligibility for nested cohort analysis:

Inclusion criteria

* Vaginal delivery at participating facility or referred to participating facility for PPH after vaginal delivery elsewhere
* Diagnosed and treated for PPH during the stepped wedge trial
* Willing and able to give informed consent
* Agree to participate in a postpartum interview before hospital discharge
* Agree to brief follow-up interview 4 weeks after delivery

Exclusion criteria

* Delivery via Cesarean section
* Transferred to another facility before delivery
* Transferred to the participating facility after vaginal delivery elsewhere but died before arrival

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60105 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Maternal death due to PPH or invasive procedures due to PPH | After delivery and before discharge from facility (usually within 48 hours after delivery)
  Proportion of women who experience maternal death due to PPH or who receive invasive procedures (including compression/B Lynch sutures, uterine artery ligation, uterine artery embolization, and hysterectomy) for PPH management. This is the primary outcome for the stepped wedge trial.
Treatment of postpartum infection among women diagnosed with PPH | Within 4 weeks after delivery
  Proportion of women diagnosed with PPH who receive antibiotics for presumptive or confirmed postpartum infection after hospital discharge and within 4 weeks postpartum. This is the primary outcome for the nested cohort analysis.

SECONDARY OUTCOMES:
Proportion of women who receive blood transfusion for PPH management | After delivery and before discharge from facility (usually within 48 hours after delivery)
  Proportion of women who receive blood transfusion for PPH management. This outcome will be assessed for the stepped wedge trial.
Transfer to next level care | After delivery and before discharge from facility (usually within 48 hours after delivery)
  Proportion of women transferred to the next level referral facility due to PPH. This outcome will be assessed for the stepped wedge trial.
Treatment for severe postpartum infection | Within 4 weeks after delivery
  Proportion of women diagnosed with PPH who are hospitalized due to postpartum infection and/or receive intravenous antibiotics to treat postpartum infection after hospital discharge and within 4 weeks postpartum. This outcome will be assessed in the nested cohort analysis.
Level of pain experienced by women postpartum | After delivery and before discharge from facility (usually within 48 hours after delivery)
  Level of pain experienced after delivery as reported by women diagnosed with PPH. Pain will be assessed using a 10-point scale. This outcome will be assessed in the nested cohort analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Anger, MPH, Principal Investigator — Gynuity Health Projects; Rasha Dabash, MPH, Principal Investigator — Gynuity Health Projects; Laura Frye, MPH, Principal Investigator — Gynuity Health Projects; Ayisha Diop, MPH, Principal Investigator — Gynuity Health Projects; Sam Ononge, MD, Principal Investigator — Makerere University; Nevine Hassanien, MD, Principal Investigator — Consultant; Mohamed Cherine Ramadan, MD, Principal Investigator — El Galaa Teaching Hospital; Emad Darwish, MD, Principal Investigator — Alexandria University; Bocar Daff, MD, Principal Investigator — Ministry of Health, Senegal; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (18):
- Egypt (6):
  - Abu Hummus Hospital, Abū Ḩummuş
  - Fayoum General Hospital, Al Fayyum
  - Ismailia General Hospital, Ismailia
  - Itsa Hospital, Iţsā
  - Etay el Barood Hospital, Ītāy al Bārūd
  - Kafr el Dawar Hospital, Kafr El Dawar
- Senegal (6):
  - Centre de Santé Gaspard Camara, Dakar
  - Centre de Santé Nabil Choucair, Dakar
  - Centre de Santé Philip Maguilene Senghor, Dakar
  - Hôpital Roi Boudoin, Dakar
  - Centre de Santé Tefess Mbour, Mbour
  - Hôpital Régional de Mbour, Mbour
- Uganda (6):
  - Gombe Hospital, Gombe
  - Itojo Hospital, Itojo
  - Kiryandongo Hospital, Kiryandongo
  - Kitagata Hospital, Kitagata
  - Lyantonde Hospital, Lyantonde
  - Masindi Hospital, Masindi

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374